CLINICAL TRIAL: NCT04338581
Title: Evaluation of AMG 714 for Vitiligo: A Phase 2a Randomized Double Blind Placebo Controlled Trial (ITN086AI)
Brief Title: Evaluation of AMG 714 for Vitiligo
Acronym: REVEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ITN086AI; NIAID CRMS ID#: 38677 (Other: DAIT NIAID)
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Vitiligo
Keywords: efficacy; facial repigmentation; randomized placebo-controlled phase 2a trial
MeSH Terms: conditions — Vitiligo | interventions — AMG-714

STUDY DESIGN:
Intervention Model Description: Phase 2a, double blind, placebo-controlled, multi-center, proof of concept trial of AMG 714 for the treatment of vitiligo. Participants will be randomized 2:1 to receive AMG 714 or placebo for AMG 714. Random assignment will be stratified by active versus stable vitiligo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMG 714 (Experimental): Participants will be administered 300 mg AMG 714 beginning at Week 0 and every 2 weeks thereafter through Week 10 (for a total of 6 doses). Each dose will be administered as 2 subcutaneous injections (1.5 mL each).
  Interventions: Biological: AMG 714; Procedure: nbUVB phototherapy
- Placebo (Placebo Comparator): Participants will be administered placebo as 2 subcutaneous injections (1.5 mL each) beginning at Week 0 and every 2 weeks thereafter through Week 10 (for a total of 6 doses).
  Interventions: Biological: Placebo; Procedure: nbUVB phototherapy

INTERVENTIONS:
Biological: AMG 714 — anti-IL-15 monoclonal antibody (Anti-IL-15 MAB)
  Arms: AMG 714
Biological: Placebo — Placebo for AMG 714
  Arms: Placebo
Procedure: nbUVB phototherapy — Participants will undergo narrow band ultraviolet B (nbUVB) phototherapy if their total body Vitiligo Area Scoring Index (T-VASI) does not improve by ≥ 25% at Week 24 compared to Week 0. Phototherapy will be administered in accordance with the Vitiligo Working Group expert recommendations.
  Other Names: narrow band ultraviolet B phototherapy

SUMMARY:
This study is designed to evaluate the efficacy of AMG 714 for the treatment of adult participants with vitiligo.

DETAILED DESCRIPTION:
The primary objective of this trial is to determine the efficacy of interleukin-15 (IL-15) inhibition with AMG 714 at inducing facial repigmentation in vitiligo.

The secondary objectives are to:

* Evaluate the safety and tolerability of AMG 714 in vitiligo
* Determine the efficacy of IL-15 inhibition with AMG 714 at inducing total body skin repigmentation in vitiligo
* Assess the durability of the skin repigmentation achieved by AMG 714 in vitiligo
* Evaluate the efficacy of AMG 714 followed by narrow band UVB (nbUVB) phototherapy

ELIGIBILITY:
Individuals must meet all of the following criteria to be eligible for enrollment as study participants:

1. Adults 18-75 years of age.
2. Clinical diagnosis of active or stable vitiligo made by a dermatologist, as defined in Protocol Section 3.4.2.
3. F-VASI ≥ 0.25 (Appendix 2 of Protocol).
4. T-VASI ≥ 3 (Appendix 2 of Protocol).
5. Willingness to:

   1. Undergo nbUVB phototherapy, as outlined in Protocol Section 7.3.
   2. Stop all other treatments for vitiligo from screening through the final follow up visit as outlined in Protocol Section 7.2.

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible for enrollment as study participants:

1. Inability or unwillingness of a participant to give written informed consent or comply with the study protocol.
2. Segmental vitiligo.
3. Contraindication to nbUVB phototherapy.
4. More than 33% leukotrichia on the face or on the total body.
5. Use of biologic immunosuppressive or immunomodulatory agents, or investigational therapy or procedure within 12 weeks or 5 half-lives prior to Visit 0 (whichever is longer), except agents authorized for prevention and treatment of SARS-CoV-2 infection according to FDA Emergency Use Authorization (EUA).
6. Use of laser or light-based treatment (phototherapy) including tanning beds within 8 weeks prior to Visit 0.
7. Use of non-biologic systemic or topical immunosuppressive or immunomodulatory agents within 4 weeks prior to Visit 0.
8. History of melanocyte-keratinocyte transplantation procedure (MKTP) or other surgical treatment for vitiligo.
9. Current or past use of the depigmenting agent monobenzyl ether of hydroquinone, including Benoquin® (Monobenzone).
10. Presence of skin conditions or lesions that would confound the vitiligo assessments.
11. Spontaneous repigmentation within 6 months prior to Visit 0 (repigmentation without any treatment and significant in amount as determined by the investigator).
12. Uncontrolled thyroid function at screening as determined by the investigator. If the participant has a history of thyroid disease and is on treatment, the participant must be on a stable thyroid regimen for at least three months prior to Visit 0.
13. Greater than 3 adequately treated nonmetastatic basal cell carcinomas (BCC) or squamous cell carcinomas (SCC) within 12 months prior to Visit 0; or previous history of multiple BCC or SCC which may pose additional risks from participation in the study in the opinion of the investigator.
14. Previous or current diagnosis of other cancer, except adequately treated cervical carcinoma in situ.
15. Acute or chronic infection, including current use of suppressive therapy for chronic infection, hospitalization for treatment of infection within 90 days prior to Visit 0, or parenteral anti-microbial (including anti-bacterial, anti-viral, or anti-fungal agents) use within 90 days prior to Visit 0.
16. Evidence of infection, including:

    1. Human immunodeficiency virus (HIV)
    2. Current or prior infection with hepatitis B (HBV), as indicated by positive HBsAg or positive HBcAb
    3. Current or prior hepatitis C (HCV), unless treated with anti-viral therapy with achievement of a sustained virologic response (undetectable viral load 12 weeks after cessation of therapy)
    4. Positive Quantiferon-TB Gold or Quantiferon-TB Gold Plus test. PPD or T-SPOT.TB test may be substituted for Quantiferon-TB Gold or Quantiferon-TB Gold Plus test
17. Any of the following laboratory abnormalities:

    1. White blood count (WBC) < 3.5 x 10^3/μL
    2. Hemoglobin < 10 g/dL
    3. Platelets (Plt) < 125,000/mm^3
    4. Alanine aminotransferase (ALT) ≥ 2x ULN
    5. Aspartate aminotransferase (AST) ≥ 2x ULN
18. Women of child-bearing potential who are unwilling to use a medically acceptable form of contraception or be sexually inactive by abstinence until study Week 48 (Protocol Section 7.4). Contraception or abstinence is required for 2 weeks prior to Visit 0.
19. Women who are pregnant or lactating.
20. Vaccination with a live attenuated vaccine within 30 days prior to Visit 0.
21. Known drug allergy or reaction to any component of AMG 714 (Protocol Section 6.1.1) or proteins derived from mammalian cell lines.
22. Past or current medical problems or findings from physical examination or laboratory testing, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
23. Current, diagnosed mental illness (e.g. severe depression) or current, diagnosed or self-reported drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett A. King, MD, PhD, Study Chair — Yale University School of Medicine: Department of Dermatology
Locations (7):
- United States (7):
  - University of California, Irvine: Department of Dermatology, Irvine, California
  - University of California Davis Health System: Department of Dermatology, Sacramento, California
  - Yale University School of Medicine: Department of Dermatology, New Haven, Connecticut
  - Tufts Medical Center: Department of Dermatology, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Northwell Health, Lake Success, New York

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access and additional relevant materials will be made available upon completion of the trial.
Time Frame: After completion of the trial, within 24 months status post database lock.
Access Criteria: The Immunology Database and Analysis Portal (ImmPort) is an open access platform for research data sharing and a long-term archive of clinical and mechanistic data, a National Institute of Allergy and Infectious Diseases Division of Allergy, Immunology and Transplantation (NIAID DAIT)-funded data repository. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort is provided by NIH-funded programs, other research organizations and individual scientists, ensuring these discoveries will be the foundation of future research.
URL: https://www.immport.org/home

REFERENCES:
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: NIH health information: Vitiligo — https://www.niams.nih.gov/health-topics/vitiligo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven sites in the United States were activated. All seven sites randomized participants. The first site was activated in November 2020 and the last participant was randomized in May 2024.
Groups:
- AMG 714: Participants receive 300 mg AMG 714 subcutaneously every 2 weeks for 6 doses beginning at Week 0 with the last dose at Week 10.
- Placebo: Participants receive placebo subcutaneously every 2 weeks for 6 doses beginning at Week 0 with the last dose at Week 10.
Period: Overall Study
Arm/Group | AMG 714 | Placebo
Started | 40 | 20 (One participant randomized but did not initiate treatment.)
Received AMG 714 | 40 | 1 (One participant received AMG 714 for their first dose and received Placebo for all subsequent doses.)
Received Placebo | 0 | 19 (One participant received AMG 714 for their first dose and received Placebo for all subsequent doses.)
Completed | 34 | 16
Not Completed | 6 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Prohibited Medication | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat (mITT) population included all randomized participants who received at least one dose of either AMG 714 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG 714 | Placebo | Total
Number analyzed (Participants) | 40 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12.75) | 52.4 (14.40) | 50.7 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 21 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 35 | 16 | 51
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 27 | 12 | 39
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 40 | 19 | 59
Vitiligo Type at Baseline [Count of Participants; unit: Participants] — Active or stable vitiligo at baseline
  Participants
    Active Vitiligo | 23 | 11 | 34
    Stable Vitiligo | 17 | 8 | 25
F-VASI at Baseline [Mean (Standard Deviation); unit: Score on a Scale] — F-VASI assesses the area of the face affected by vitiligo. F-VASI is determined by the product of the percent of vitiligo involvement (percent of body surface area [BSA]) and the degree of depigmentation estimated to the nearest of the following percentages: 0%, 10%, 25%, 50%, 75%, 90%, or 100%. The percentage of BSA (hand or thumb unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator. F-VASI has a possible range from 0 to 3.5, with higher scores indicating more severe disease.
  Score on a Scale | 1.154 (0.8982) | 1.035 (0.9513) | 1.116 (0.9091)
T-VASI at Baseline [Mean (Standard Deviation); unit: Score on a Scale] — T-VASI assesses the area of the body affected by vitiligo. The body is divided into 6 regions: head and neck, upper extremities, hands, torso, lower extremities, and feet. For each body region, the VASI is determined by the product of the percent of vitiligo involvement (percent of body surface area [BSA]) and the degree of depigmentation estimated to the nearest of the following percentages: 0%, 10%, 25%, 50%, 75%, 90%, or 100%. T-VASI is derived by summing the values of all body regions, providing a possible range from 0 to 99, with higher scores indicating more severe disease.
  Score on a Scale | 19.901 (21.4012) | 18.884 (15.0015) | 19.573 (19.4434)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving a ≥ 35% Improvement From Baseline in the Facial Vitiligo Area Scoring Index (F-VASI35) at Week 24
Description: An F-VASI35 responder is defined as a participant who has at least 35% improvement from Baseline in the facial vitiligo area scoring index (F-VASI). F-VASI assesses the area of the face affected by vitiligo. F-VASI is determined by the product of the percent of vitiligo involvement (percent of body surface area [BSA]) and the degree of depigmentation estimated to the nearest of the following percentages: 0%, 10%, 25%, 50%, 75%, 90%, or 100%. The percentage of BSA (hand or thumb unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator. F-VASI has a possible range from 0 to 3.5, with higher scores indicating more severe disease. Participants missing the F-VASI assessment at Week 24 are imputed as F-VASI35 non-responders.
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 40 | 19
Proportion of participants | 0.150 [0.057 to 0.298] | 0.053 [0.001 to 0.260]
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; The p-value compares AMG 714 and Placebo treatment groups; Test type: Superiority; p = 0.411, Fisher Exact — P-value is from comparing the proportion of F-VASI35 Responders between the two treatment groups using a Fisher's exact test

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were recorded in EDC from after treatment initiation at Week 0 to Week 48.
Description: Generalized pruritus or urticaria Grade 1 hypersensitivity/anaphylaxis reactions, confirmed Grade 1 SARS-CoV-2 infections, and Grade 2 or higher AEs were recorded in EDC. Safety analyses are based on the safety population, which consists of all participants who receive any amount of AMG 714 or placebo. Participants will be analyzed according to the actual treatment received. One participant randomized to the placebo group received AMG 714.
Groups:
- AMG 714: Participants receive 300 mg AMG 714 subcutaneously every 2 weeks for 6 doses beginning at Week 0 with the last dose at Week 10. Any participant receiving at least one injection of AMG 714 at any time during the study will be summarized with the AMG 714 treatment arm.
Arm/Group | AMG 714 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/18
Other Adverse Events (participants affected / at risk) | 23/41 | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMG 714 (N=41) | Placebo (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT04338581/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04338581/ICF_001.pdf